CLINICAL TRIAL: NCT02940860
Title: A Phase III, Randomised, Open-label, Comparative Safety and Efficacy Trial of Intravenous Iron Isomaltoside/Ferric Derisomaltose (Monofer®/Monoferric®) and Iron Sucrose in Subjects With Iron Deficiency Anaemia and Non-dialysis-dependent Chronic Kidney Disease (FERWON-NEPHRO)
Brief Title: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose for Treatment of Iron Deficiency Anemia in Non-Dialysis-Dependent Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-CKD-04
Record Dates: First submitted 2016-09-27; First posted 2016-10-21 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-02

CONDITIONS: Iron Deficiency Anaemia; Iron Deficiency Anemia; Chronic Kidney Disease
Keywords: Iron Deficiency Anaemia; Iron Deficiency Anemia; IDA; Chronic Kidney Disease; CKD; Iron isomaltoside; Ferric derisomaltose; Monofer; Monoferric; Monover; Monofar; Monoferro
MeSH Terms: conditions — Anemia, Iron-Deficiency; Renal Insufficiency, Chronic | interventions — iron isomaltoside 1000; ferric derisomaltose; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron isomaltoside/ferric derisomaltose (Experimental): Administered IV
  Interventions: Drug: Iron isomaltoside/ferric derisomaltose
- Iron sucrose (Active Comparator): Administered IV
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Iron isomaltoside/ferric derisomaltose — Iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) was the test product in this trial.
  The dose of iron isomaltoside/ferric derisomaltose for the individual subject was set to 1000 mg. The dose was diluted in 100 mL 0.9 % sodium chloride (100 mL bags) and administered as a single IV infusion over approximately 20 minutes.
  Other Names: Monofer®, Monoferric®, Monover®, Monofar®, Monoferro®
  Arms: Iron isomaltoside/ferric derisomaltose
Drug: Iron sucrose — Iron sucrose (Venofer®; 20 mg elemental iron/mL) was the comparator in this trial. Iron sucrose was administered as 200 mg undiluted IV injections over approximately 2-5 minutes and repeated according to standard practice or physician choice up to a maximum of five times within the first two weeks starting at baseline. A cumulative dose of 1000 mg was recommended.
  Other Names: Venofer®
  Arms: Iron sucrose

SUMMARY:
Evaluation of safety and efficacy of iron isomaltoside/ferric derisomaltose compared with iron sucrose, in subjects with both non-dialysis-dependent chronic kidney disease (NDD-CKD) and iron deficiency anaemia (IDA).

DETAILED DESCRIPTION:
Iron deficiency anaemia (IDA) is a common problem associated with many chronic diseases such as chronic kidney disease (CKD). IDA can have a substantial medical and quality of life (QoL) burden on the subjects. Therapy of these subjects includes treating the underlying cause of IDA and restoring haemoglobin (Hb) concentration and iron stores.

This study evaluated the safety and efficacy of iron isomaltoside/ferric derisomaltose compared with iron sucrose in subjects with both non-dialysis-dependent chronic kidney disease (NDD-CKD) and iron deficiency anaemia (IDA).

The study subjects received either a single intravenous (IV) dose of iron isomaltoside/ferric derisomaltose (1000 mg at baseline) or iron sucrose (200 mg IV injections at baseline and repeated according to standard practice or physician choice up to a maximum of five times within the first two weeks starting at baseline; a cumulative dose of 1000 mg was recommended). The study subjects were monitored for up to 8 weeks from baseline.

ELIGIBILITY:
Inclusion Criteria includes:

1. Men and women, ≥ 18 years
2. Hb ≤ 11 g/dL
3. Chronic renal impairment, as defined by either (i) eGFR < 60 mL/min/1.73m2 at screening (as calculated by modification of diet in renal disease (MDRD)), or (ii) Estimated Glomerular Filtration Rate (eGFR) < 90 mL/min/1.73m2 at screening and kidney damage as indicated by abnormalities in urine composition per medical history and/or intermediate/high risk of cardio-vascular disease based on the Framingham model
4. Screening s-ferritin ≤ 100 ng/mL, or ≤ 300 ng/mL if Transferrin Saturation (TSAT) ≤ 30 %
5. Either no Erythropoiesis Stimulating Agent (ESAs) or ESAs as a stable dose 4 weeks before randomisation
6. Willingness to participate and signing the informed consent form

Exclusion Criteria includes:

1. Anaemia predominantly caused by factors other than IDA
2. Hemochromatosis or other iron storage disorders
3. Previous serious hypersensitivity reactions to any IV iron compounds
4. Prior to screening or during the trial period; has or will be treated with a red blood cell transfusion, radiotherapy, and/or chemotherapy
5. Undergoing dialysis for treatment of CKD
6. Planned surgical procedure within the trial period
7. Decompensated liver cirrhosis or active hepatitis
8. Alcohol or drug abuse within the past 6 month.
9. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1538 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacosmos A/S Clinical and Non-clinical Research, Study Director — Pharmacosmos A/S
Locations (112):
- United States (112):
  - Pharmacosmos Investigational Site, Huntsville, Alabama
  - Pharmacosmos Investigational Site, Little Rock, Arkansas
  - Pharmacosmos Investigational Site, Chula Vista, California
  - Pharmacosmos Investigational Site, Fresno, California
  - Pharmacosmos Investigational Site, Glendale, California
  - Pharmacosmos Investigational Site, Granada Hills, California
  - Pharmacosmos Investigational Site, La Mesa, California
  - Pharmacosmos Investigational Site, Los Angeles, California
  - Pharmacosmos Investigational Site1, Los Angeles, California
  - Pharmacosmos Investigational Site2, Los Angeles, California
  - Pharmacosmos Investigational Site, Lynwood, California
  - Pharmacosmos Investigational Site, Montebello, California
  - Pharmacosmos Investigational Site, Northridge, California
  - Pharmacosmos Investigational Site, Porterville, California
  - Pharmacosmos Investigational Site, Rialto, California
  - Pharmacosmos Investigational Site, Riverside, California
  - Pharmacosmos Investigational Site, Sacramento, California
  - Pharmacosmos Investigational Site, San Dimas, California
  - Pharmacosmos Investigational Site, San Francisco, California
  - Pharmacosmos Investigational Site, Tarzana, California
  - Pharmacosmos Investigational Site, Arvada, Colorado
  - Pharmacosmos Investigational Site, Denver, Colorado
  - Pharmacosmos Investigational Site, Westminster, Colorado
  - Pharmacosmos Investigational Site, Middlebury, Connecticut
  - Pharmacosmos Investigational Site, Plainville, Connecticut
  - Pharmacosmos Investigational Site, Boynton Beach, Florida
  - Pharmacosmos Investigational Site, Brandon, Florida
  - Pharmacosmos Investigational Site, Coral Gables, Florida
  - Pharmacosmos Investigational Site, Coral Springs, Florida
  - Pharmacosmos Investigational Site, Doral, Florida
  - Pharmacosmos Investigational Site, Fort Lauderdale, Florida
  - Pharmacosmos Investigational Site1, Hialeah, Florida
  - Pharmacosmos Investigational Site2, Hialeah, Florida
  - Pharmacosmos Investigational Site3, Hialeah, Florida
  - Pharmacosmos Investigational Site, Hollywood, Florida
  - Pharmacosmos Investigational Site, Homestead, Florida
  - Pharmacosmos Investigational Site, Lake City, Florida
  - Pharmacosmos Investigational Site1, Lauderdale Lakes, Florida
  - Pharmacosmos Investigational Site2, Lauderdale Lakes, Florida
  - Pharmacosmos Investigational Site1, Miami, Florida
  - Pharmacosmos Investigational Site2, Miami, Florida
  - Pharmacosmos Investigational Site, Miami, Florida
  - Pharmacosmos Investigational Site3, Miami, Florida
  - Pharmacosmos Investigational Site, Miami Beach, Florida
  - Pharmacosmos Investigational Site, Miami Lakes, Florida
  - Pharmacosmos Investigational Site, Naples, Florida
  - Pharmacosmos Investigational Site, Ocala, Florida
  - Pharmacosmos Investigational Site, Palmetto Bay, Florida
  - Pharmacosmos Investigational Site, Pembroke Pines, Florida
  - Pharmacosmos Investigational Site, Plantation, Florida
  - Pharmacosmos Investigational Site, Port Charlotte, Florida
  - Pharmacosmos Investigational Site, St. Petersburg, Florida
  - Pharmacosmos Investigational Site1, Tampa, Florida
  - Pharmacosmos Investigational Site2, Tampa, Florida
  - Pharmacosmos Investigational Site, Tampa, Florida
  - Pharmacosmos Investigational Site, West Miami, Florida
  - Pharmacosmos Investigational Site, Atlanta, Georgia
  - Pharmacosmos Investigational Site, Augusta, Georgia
  - Pharmacosmos Investigational Site, Macon, Georgia
  - Pharmacosmos Investigational Site, Chicago, Illinois
  - Pharmacosmos Investigational Site, Crystal Lake, Illinois
  - Pharmacosmos Investigational Site, Hinsdale, Illinois
  - Pharmacosmos Investigational Site, Fort Wayne, Indiana
  - Pharmacosmos Investigational Site, Marion, Indiana
  - Pharmacosmos Investigational Site, Merrillville, Indiana
  - Pharmacosmos Investigational Site, Michigan City, Indiana
  - Pharmacosmos Investigational Site, Kansas City, Kansas
  - Pharmacosmos Investigational Site, Wichita, Kansas
  - Pharmacosmos Investigational Site, Owensboro, Kentucky
  - Pharmacosmos Investigational Site, Baton Rouge, Louisiana
  - Pharmacosmos Investigational Site, Covington, Louisiana
  - Pharmacosmos Investigational Site, Shreveport, Louisiana
  - Pharmacosmos Investigational Site, Annapolis, Maryland
  - Pharmacosmos Investigational Site, Bethesda, Maryland
  - Pharmacosmos Investigational Site, Rockville, Maryland
  - Pharmacosmos Investigational Site, Grand Rapids, Michigan
  - Pharmacosmos Investigational Site, Florissant, Missouri
  - Pharmacosmos Investigational Site, Albuquerque, New Mexico
  - Pharmacosmos Investigational Site, Flushing, New York
  - Pharmacosmos Investigational Site, New York, New York
  - Pharmacosmos Investigational Site, Asheville, North Carolina
  - Pharmacosmos Investigational Site, Gastonia, North Carolina
  - Pharmacosmos Investigational Site, Greenville, North Carolina
  - Pharmacosmos Investigational Site, Jacksonville, North Carolina
  - Pharmacosmos Investigational Site, Wilmington, North Carolina
  - Pharmacosmos Investigational Site, Cincinnati, Ohio
  - Pharmacosmos Investigational Site, Cleveland, Ohio
  - Pharmacosmos Investigational Site, Norman, Oklahoma
  - Pharmacosmos Investigational Site, Tulsa, Oklahoma
  - Pharmacosmos Investigational Site, Bethlehem, Pennsylvania
  - Pharmacosmos Investigational Site, Philadelphia, Pennsylvania
  - Pharmacosmos Investigational Site, Columbia, South Carolina
  - Pharmacosmos Investigational Site, Greenville, South Carolina
  - Pharmacosmos Investigational Site, Orangeburg, South Carolina
  - Pharmacosmos Investigational Site, Jackson, Tennessee
  - Pharmacosmos Investigational Site, Austin, Texas
  - Pharmacosmos Investigational Site, Beaumont, Texas
  - Pharmacosmos Investigational Site, DeSoto, Texas
  - Pharmacosmos Investigational Site, El Paso, Texas
  - Pharmacosmos Investigational Site, Fort Worth, Texas
  - Pharmacosmos Investigational Site, Greenville, Texas
  - Pharmacosmos Investigational Site1, Houston, Texas
  - Pharmacosmos Investigational Site2, Houston, Texas
  - Pharmacosmos Investigational Site, Houston, Texas
  - Pharmacosmos Investigational Site, Lufkin, Texas
  - Pharmacosmos Investigational Site, McKinney, Texas
  - Pharmacosmos Investigational Site, Pearland, Texas
  - Pharmacosmos Investigational Site1, San Antonio, Texas
  - Pharmacosmos Investigational Site2, San Antonio, Texas
  - Pharmacosmos Investigational Site, St. George, Utah
  - Pharmacosmos Investigational Site, Arlington, Virginia
  - Pharmacosmos Investigational Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sunil Bhandari, Lars Lykke Thomsen. Single 1000 mg infusion of iron isomaltoside1000 single 1000 mg infusion of iron isomaltoside 1000 demonstrates a more rapid hemoglobin response and reduced risk of cardiovascular adverse events compared to multiple dose iron sucrose In patients with iron deficiency anemia and nondialysis-dependent CKD. Nephrology Dialysis Transplantation 34 (Supplement 1): i349-i350, 2019, https://academic.oup.com/ndt/article/34/Supplement_1/gfz101.SaO035/5515662
- [Derived] Bhandari S, Kalra PA, Berkowitz M, Belo D, Thomsen LL, Wolf M. Safety and efficacy of iron isomaltoside 1000/ferric derisomaltose versus iron sucrose in patients with chronic kidney disease: the FERWON-NEPHRO randomized, open-label, comparative trial. Nephrol Dial Transplant. 2021 Jan 1;36(1):111-120. doi: 10.1093/ndt/gfaa011. PMID 32049331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2560 subjects were screened and 1538 subjects were randomised into the trial.
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) was the test product in this trial.
  Subjects received iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) as a single IV infusion of 1000 mg at the baseline visit.
- Iron Sucrose: Iron sucrose (Venofer®) was the comparator in this trial.
  Subjects received iron sucrose (Venofer®), 200 mg IV injection up to a maximum of 5 IV injections within the first 2 weeks, starting at baseline (a cumulative dose of 1000 mg was recommended).
Period: Overall Study
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Started | 1027 | 511
Completed | 971 | 476
Not Completed | 56 | 35
Not completed — Non-serious AE | 1 | 2
Not completed — Serious AE | 7 | 3
Not completed — Withdrawal by Subject | 19 | 9
Not completed — Lost to Follow-up | 13 | 7
Not completed — Physician Decision | 5 | 3
Not completed — Sponsor Decision | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Death | 3 | 2
Not completed — Moved, poor venous access, transport | 6 | 4
Not completed — Not treated | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Iron isomaltoside/ferric derisomaltose, administered IV
- Iron Sucrose: Iron sucrose, administered IV
- Total: Total of all reporting groups
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose | Total
Number analyzed (Participants) | 1027 | 511 | 1538
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (12.3) | 69.3 (12.3) | 68.6 (12.3)
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 337 | 151 | 488
  65-84 years | 608 | 316 | 924
  > 84 years | 82 | 44 | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 633 | 329 | 962
  Male | 394 | 182 | 576
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 476 | 248 | 724
  Not Hispanic or Latino | 551 | 263 | 814
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 16 | 11 | 27
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 264 | 117 | 381
  White | 731 | 375 | 1106
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 11 | 6 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Mexican | 4 | 3 | 7
  Indigenous Mexican | 1 | 0 | 1
  Mixed (Caucasian and Native american) | 1 | 0 | 1
  Hispanic | 4 | 3 | 7
  Central Indian | 1 | 0 | 1
  Guyanese | 1 | 0 | 1
  Other (Mixed: not declared) | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1027 | 511 | 1538
Current smoker [Number; unit: participants]
  YES | 118 | 53 | 171
  NO | 909 | 458 | 1367

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hb) From Baseline to Week 8
Description: Efficacy
  Evaluate the effect of iron isomaltoside/ferric derisomaltose vs iron sucrose in subjects with non-dialysis-dependent chronic kidney disease (NDD-CKD) and iron deficiency anaemia (IDA).
  Response was defined as change from baseline in hemoglobin (Hb) to week 8, i.e. ability to increase Hb in subjects with NDD-CKD and IDA, when oral iron preparations were ineffective or could not be used, or in whom the Hb measurement at screening in Investigators' opinion were sufficiently low to require rapid repletion of iron stores.
Time Frame: Baseline to week 8
Population: Intention to treat (ITT). All randomised subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
g/dL | 1.22 [1.14 to 1.31] | 1.14 [1.03 to 1.26]
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Power: With N=1000 subjects in the iron isomaltoside/ferric derisomaltose treatment group and with N=500 subjects in the iron sucrose treatment group, assuming no difference between the treatment groups and assuming a common standard deviation (SD) of 1.5 g/dL, the power was 100% for demonstrating non-inferiority of the change in Hb from baseline to week 8, using a non-inferiority margin of -0.5 g/dL. The significance level was set to 5%; Test type: Non-Inferiority — Non-inferiority could be claimed if the lower bound of the 95% confidence interval (CI) was above -0.5 g/dL; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.06 to 0.23] — The Mixed Model for Repeated Measurement (MMRM) used for testing, included the fixed, categorical effects of treatment, week, treatment-by-week interaction, strata, and the continuous covariates of baseline Hb and baseline Hb-by-week interaction

2. Primary Outcome: Incidence of Protocol-defined Serious or Severe Hypersensitivity Reactions
Description: Safety
  For this endpoint, the number of participants with serious or severe hypersensitivity reactions were evaluated. The hypersensitivity reactions that were included in the analysis were those that started on or after the first dose of randomised treatment (i.e. treatment emergent). The terms used to define hypersensitivity were those specified by the Standardised MedDRA Queries (SMQ) for hypersensitivity, plus four additional terms: loss of consciousness, seizure, syncope, unresponsiveness.
  The potential hypersensitivity AEs were adjudicated in a blinded fashion by an independent Clinical Endpoint Adjudication Committee (CEAC).
  Results show only those participants that had adjudicated and confirmed serious or severe hypersensitivity reactions.
Time Frame: Baseline to week 8
Population: Safety analysis set. All randomised subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1019 | 506
Participants | 3 | 0
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose; Power: With N=1000 subjects in the iron isomaltoside/ferric derisomaltose, the power was 88% to demonstrate that the upper bound of the 95% CI of the incidence of treatment-emergent serious and/or severe non-serious hypersensitivity AEs was less than 3%. The significance level was set to 5%; Test type: Other; 95% two-sided CI (iron isomaltoside) = 0.3, 95% CI 2-sided [0.06 to 0.86]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Risk difference between iron isomaltoside/ferric derisomaltose and iron sucrose was assessed for the individual trial with 95% Newcombe CI adjusted for stratum using the Cochran-Mantel-Haenszel method; Test type: Other; Risk Difference (RD) = 0.29, 95% CI 2-sided [-0.19 to 0.77]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Risk difference between iron isomaltoside/ferric derisomaltose and iron sucrose was assessed for the pooled FERWON-IDA and FERWON-NEPHRO trials (2008 subjects treated with iron isomaltoside/ferric derisomaltose and 1000 subjects treated with iron sucrose) with 95% Newcombe CI adjusted for stratum using the Cochran-Mantel-Haenszel method; Test type: Non-Inferiority — Non-inferiority can be claimed if the upper bound of the 95% CI is below 1.5 % point; Risk Difference (RD) = 0.10, 95% CI 2-sided [-0.57 to 0.48]

3. Secondary Outcome: Composite Cardiovascular Adverse Events (AEs)
Description: Safety
  Results show the composite cardiovascular AEs, that started on or after the first dose of randomised treatment (i.e. treatment emergent) up to week 8.
  The reported potential cardiovascular AEs were adjudicated in a blinded fashion by an independent Clinical Endpoint Adjudication Committee (CEAC).
  The potential cardiovascular AEs included the following:
  * Death due to any cause
  * Non-fatal myocardial infarction
  * Non-fatal stroke
  * Unstable angina requiring hospitalisation
  * Congestive heart failure requiring hospitalisation or medical intervention
  * Arrhythmias
  * Hypertension
  * Hypotension
  Results show only those participants that had adjudicated and confirmed treatment-emergent composite cardiovascular AEs.
Time Frame: Baseline, week 1, 2, and 8
Population: Safety analysis set. All randomised subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1019 | 506
Participants | 42 | 35
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Adjudicated and confirmed treatment-emergent composite cardiovascular AEs. Any treatment emergent composite cardiovascular AEs were included in the statistical evaluation. The overall incidence of adjudicated and confirmed composite cardiovascular AEs was tabulated and compared between the treatment groups by a Fisher's exact test; Test type: Superiority; p = 0.0248, Fisher Exact

4. Secondary Outcome: Time to First Composite Cardiovascular Safety AE
Description: Safety
  Time to first composite cardiovascular AE was defined as the actual time in days from first dose of treatment until the date of the composite cardiovascular AE. For subjects not reporting a composite cardiovascular AE, the time was censored at the date of the last attended visit. Only the adjudicated and confirmed composite cardiovascular safety AEs, as judged by the CEAC, were considered for this endpoint.
  Time to first composite cardiovascular AE was defined as the actual time in days from first dose of treatment until the date of the composite cardiovascular AE. For subjects not reporting a composite cardiovascular AE, the time was censored at the date of the last attended visit.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: Safety analysis set. All randomised subjects who received at least one dose of the investigational product.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1019 | 506
Week | NA [NA to NA] — The number of adjudicated and confirmed composite cardiovascular safety AEs was too low (N=42) for estimation of median and 95% CI. | NA [NA to NA] — The number of adjudicated and confirmed composite cardiovascular safety AEs was too low (N=35) for estimation of median and 95% CI.
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; The time to first adjudicated and confirmed composite cardiovascular AEs was estimated using the Kaplan-Meier method and the hypothesis of no treatment difference was assessed by a log-rank test; Test type: Superiority; p = 0.0185, Log Rank

5. Secondary Outcome: S-phosphate <2 mg/dL at Any Time From Baseline to Week 1, 2, 4, and 8
Description: Safety
  Results show the number of participants who had s-phosphate <2 mg/dL at any time from baseline to week 1, 2, 4, or 8.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: Safety analysis set. All randomised subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1011 | 500
Participants | 32 | 4

6. Secondary Outcome: Hb Concentration Increase of ≥1 g/dL From Baseline to Week 1, 2, 4, and 8
Description: Efficacy
  Results show Hb responders to the treatment. A subject was considered a Hb responder to a certain week if an increase in Hb of at least 1 g/dL from baseline to the week in question was observed (from baseline to week 1, 2, 4, and 8).
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
Participants
  Responder YES week 1: number analyzed (Participants) | 1002 | 494
  Responder YES week 1 | 200 | 78
  Responder YES week 2: number analyzed (Participants) | 980 | 474
  Responder YES week 2 | 339 | 112
  Responder YES week 4: number analyzed (Participants) | 957 | 469
  Responder YES week 4 | 430 | 174
  Responder YES week 8: number analyzed (Participants) | 967 | 475
  Responder YES week 8 | 474 | 226
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Hb increase of ≥1 g/dL from baseline to week 1. Proportion of Hb responders to each week was analysed using a repeated measures logistic regression model with treatment, visit, strata, and treatment by visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0478, Repeated measures logistic regressioin; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.00 to 1.87]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Hb increase of ≥1 g/dL from baseline to week 2. Proportion of Hb responders to each week was analysed using a repeated measures logistic regression model with treatment, visit, strata, and treatment by visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p < 0.0001, Repeated measures logistic regressioin; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.39 to 2.36]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Hb increase of ≥1 g/dL from baseline to week 4. Proportion of Hb responders to each week was analysed using a repeated measures logistic regression model with treatment, visit, strata, and treatment by visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0048, Repeated measures logistic regressioin; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.11 to 1.79]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Hb increase of ≥1 g/dL from baseline to week 8. Proportion of Hb responders to each week was analysed using a repeated measures logistic regression model with treatment, visit, strata, and treatment by visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.9440, Repeated measures logistic regressioin; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.80 to 1.27]

7. Secondary Outcome: Time to Change in Hb Concentration ≥1 g/dL
Description: Efficacy
  Time to change in Hb concentration ≥1 g/dL.
  Subjects who showed Hb concentration increase of ≥1 g/dL (from baseline to week 1, 2, 4, and 8).
  For responders, time to Hb response was defined as the scheduled time from baseline until the visit where the first Hb response was measured.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
Days | 56 [28 to 56] | 56 [28 to NA] — The 95% Confidence Interval value for this treatment group could not be calculated.
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Time to Hb response was estimated using the Kaplan-Meier method and the hypothesis of no treatment difference was assessed by a 2-sided log-rank test; Test type: Superiority; p = 0.0174, Log Rank

8. Secondary Outcome: Hb Concentration of >12 g/dL at Any Time From Week 1 to Week 8
Description: Efficacy
  Hb concentration of >12 g/dL at any time from week 1 to week 8.
  Results show the number of participants who achieved Hb concentration of >12 g/dL at any time from week 1 to week 8.
Time Frame: Week 1 to week 8
Population: ITT. All randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 510
Participants | 259 | 121
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; The proportion of subjects who achieved a Hb level of >12 g/dL at any time from week 1 to week 8 was analysed using a logistic regression model with treatment and strata as fixed effects. The estimated treatment ratio of iron isomaltoside/ferric derisomaltose versus iron sucrose is presented with 95% CI and corresponding p-value; Test type: Superiority; p = 0.5074, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.83 to 1.45]

9. Secondary Outcome: Hb Concentration Increase of ≥2 g/dL at Any Time From Week 1 to Week 8
Description: Efficacy
  Results show the number of participants who achieved Hb concentration increase of ≥2 g/dL at any time from week 1 to week 8.
Time Frame: Week 1 to week 8
Population: ITT. All randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 510
Participants | 307 | 133
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; The proportion of subjects who achieved an increase in Hb concentration ≥2 g/dL at any time from week 1 to week 8 was analysed using a logistic regression model with treatment and strata as fixed effects. The estimated treatment ratio of iron isomaltoside/ferric derisomaltose versus iron sucrose was presented with 95% CI and corresponding p-value; Test type: Superiority; p = 0.1035, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.96 to 1.60]

10. Secondary Outcome: S-Ferritin Concentration of ≥100 ng/mL and Transferrin Saturation (TSAT) of 20-50% at Any Time From Week 1 to Week 8
Description: Efficacy
  Proportion of subjects reaching the composite endpoint of s-ferritin concentration ≥100 ng/mL and TSAT of 20-50% at any time from week 1 to 8.
Time Frame: Week 1 to week 8
Population: ITT. All randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1012 | 500
Participants | 873 | 388
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Proportion of subject who achieved a s-ferritin level of ≥100 ng/mL AND a TSAT of 20-50% at any time from week 1 to week 8 was analysed using a logistic regression model with treatment and strata as fixed effects. The estimated treatment ratio of iron isomaltoside/ferric derisomaltose versus iron sucrose is presented with 95% CI and corresponding p-value; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.38 to 2.40]

11. Secondary Outcome: Change in Hb Concentration From Baseline to Week 1, 2, and 4
Description: Efficacy
  Change in Hb concentration from baseline to week 1, 2, and 4.
Time Frame: Baseline, week 1, 2, and 4
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
g/dL
  Week 1: number analyzed (Participants) | 1001 | 494
  Week 1 | 0.44 (0.94) | 0.21 (1.02)
  Week 2: number analyzed (Participants) | 980 | 474
  Week 2 | 0.77 (1.16) | 0.50 (1.15)
  Week 4: number analyzed (Participants) | 957 | 469
  Week 4 | 1.08 (1.32) | 0.90 (1.33)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in Hb concentration from baseline to week 1 was analysed using a MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [0.12 to 0.31]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in Hb concentration from baseline to week 2 was analysed using a MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.14 to 0.36]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Change in Hb concentration from baseline to week 4 was analysed using a MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates; Test type: Superiority; p = 0.0208, Mixed model for repeated measures; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.02 to 0.28]

12. Secondary Outcome: Change in S-ferritin From Baseline to Weeks 1, 2, 4, and 8
Description: Efficacy
  Changes in s-ferritin from baseline to weeks 1, 2, 4, and 8.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
ng/mL
  Week 1: number analyzed (Participants) | 991 | 485
  Week 1 | 492.4 (309.7) | 183.9 (129.4)
  Week 2: number analyzed (Participants) | 994 | 476
  Week 2 | 381.2 (283.8) | 292.4 (210.4)
  Week 4: number analyzed (Participants) | 968 | 472
  Week 4 | 258.4 (214.5) | 255.4 (265.6)
  Week 8: number analyzed (Participants) | 973 | 480
  Week 8 | 191.3 (196.1) | 187.9 (210.6)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in concentrations of s-ferritin from baseline to week 1 was analysed using a MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 309.2, 95% CI 2-sided [280.7 to 337.8]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in concentrations of s-ferritin from baseline to week 2 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 95.8, 95% CI 2-sided [67.9 to 123.7]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Change in concentrations of s-ferritin from baseline to week 4 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.7834, Mixed model for repeated measures; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-21.2 to 28.1]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Change in concentrations of s-ferritin from baseline to week 8 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.7621, Mixed model for repeated measures; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-18.1 to 24.7]

13. Secondary Outcome: Change in Transferrin Saturation (TSAT) From Baseline to Week 1, 2, 4, and 8
Description: Efficacy
  Changes in transferrin saturation (TSAT) from baseline to week 1, 2, 4, and 8.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
percent
  Week 1: number analyzed (Participants) | 989 | 478
  Week 1 | 12.10 (31.99) | 4.31 (23.10)
  Week 2: number analyzed (Participants) | 989 | 471
  Week 2 | 5.84 (29.79) | 5.64 (14.35)
  Week 4: number analyzed (Participants) | 964 | 472
  Week 4 | 4.99 (30.00) | 5.59 (12.31)
  Week 8: number analyzed (Participants) | 969 | 477
  Week 8 | 5.10 (30.17) | 5.93 (12.86)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in TSAT from baseline to week 1 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 8.8, 95% CI 2-sided [6.9 to 10.7]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in TSAT from baseline to week 2 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.0129, Mixed model for repeated measures; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.3 to 2.4]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Change in TSAT from baseline to week 4 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.2403, Mixed model for repeated measures; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.4 to 1.5]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Change in TSAT from baseline to week 8 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.8094, Mixed model for repeated measures; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.9 to 1.2]

14. Secondary Outcome: Change in Concentration of S-iron From Baseline to Week 1, 2, 4, and 8
Description: Efficacy
  Changes in the concentrations of serum iron (s-iron) from baseline to week 1, 2, 4, and 8.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
μg/dL
  Week 1: number analyzed (Participants) | 940 | 458
  Week 1 | 34.8 (99.7) | 11.1 (71.1)
  Week 2: number analyzed (Participants) | 938 | 449
  Week 2 | 11.1 (90.6) | 12.4 (44.1)
  Week 4: number analyzed (Participants) | 917 | 447
  Week 4 | 6.5 (91.2) | 10.2 (38.3)
  Week 8: number analyzed (Participants) | 925 | 451
  Week 8 | 7.1 (91.3) | 12.4 (41.9)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in s-iron from baseline to week 1 was analysed using a Mixed Model for Repeated Measurement (MMRM) including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by week interaction effects are presented by week, including 95% CIs and corresponding p-value; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 26.5, 95% CI 2-sided [20.4 to 32.7]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in s-iron from baseline to week 2 was analysed using a Mixed Model for Repeated Measurement (MMRM) including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by week interaction effects are presented by week, including 95% CIs and corresponding p-value; Test type: Superiority; p = 0.2229, Mixed model for repeated measures; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-1.2 to 5.1]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Change in s-iron from baseline to week 4 was analysed using a Mixed Model for Repeated Measurement (MMRM) including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by week interaction effects are presented by week, including 95% CIs and corresponding p-value; Test type: Superiority; p = 0.9046, Mixed model for repeated measures; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.9 to 2.6]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Change in s-iron from baseline to week 8 was analysed using a Mixed Model for Repeated Measurement (MMRM) including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by week interaction effects are presented by week, including 95% CIs and corresponding p-value; Test type: Superiority; p = 0.1307, Mixed model for repeated measures; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-5.8 to 0.8]

15. Secondary Outcome: Change in Fatigue Symptoms From Baseline to Week 1, 2, and 8
Description: Efficacy
  Change in fatigue symptoms from baseline to week 1, 2, and 8 was measured by the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale.
  The Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale consisted of 13 items ranging from 0 (not at all) to 4 (very much), except items #7 and #8 which are reversed scored. The total score range is 0-52.
  A score of less than 30 indicated severe fatigue, and the higher the score, the better outcome/quality of life (QoL). If more than 50% of the items for a subject at a given visit were missing, the total score was not calculated.
  Total score was calculated as shown below:
  Total score= Sum of individual scores x 13 / Number of items answered
Time Frame: Baseline, week 1, 2, and 8
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
score on a scale
  Week 1: number analyzed (Participants) | 995 | 492
  Week 1 | 5.04 (8.85) | 5.01 (7.93)
  Week 2: number analyzed (Participants) | 998 | 482
  Week 2 | 7.29 (9.84) | 7.63 (9.74)
  Week 8: number analyzed (Participants) | 976 | 483
  Week 8 | 9.13 (11.09) | 9.07 (11.40)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in fatigue symptoms score from baseline to week 1 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline score and baseline score-by-week interaction as covariates; Test type: Superiority; p = 0.8196, Mixed model for repeated measures; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.73 to 0.92]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in fatigue symptoms score from baseline to week 2 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline score and baseline score-by-week interaction as covariates; Test type: Superiority; p = 0.7132, Mixed model for repeated measures; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-1.06 to 0.73]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Change in fatigue symptoms score from baseline to week 8 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline score and baseline score-by-week interaction as covariates; Test type: Superiority; p = 0.5860, Mixed model for repeated measures; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.71 to 1.25]

16. Secondary Outcome: Intervals in Screening for Diabetic Retinopathy (ISDR) Questionnaire, Cost of Public Transport/Taxi And Parking
Description: Pharmacoeconomics
  The Intervals in Screening for Diabetic Retinopathy (ISDR) questionnaire at the baseline visit assessed the resources used by subjects to receive treatment. Resources used on other trial activities were not included. ISDR responses were summarised using descriptive statistics.
  The data for this endpoint show the responses at baseline for both treatment groups.
  The frequency of drug administration between the 2 treatment groups is different, however, (i.e. up to a factor 5 in the iron sucrose treatment group).
Time Frame: Baseline
Population: ITT. All randomised subjects.
Measure: Median (Full Range); unit: US dollars ($)
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
US dollars ($)
  Cost of public transport/taxi: number analyzed (Participants) | 131 | 57
  Cost of public transport/taxi | 0.0 [0 to 87] | 0.0 [0 to 46]
  Cost of parking: number analyzed (Participants) | 879 | 447
  Cost of parking | 0.0 [0 to 45] | 0.0 [0 to 25]

17. Secondary Outcome: Intervals in Screening for Diabetic Retinopathy (ISDR) Questionnaire, Return Journey by Car
Description: as for outcome 16
Time Frame: Baseline
Population: ITT. All randomised subjects. The number of participants analyzed were less the number of participants starting the study since not all participants had data collected for this outcome measure.
Measure: Median (Full Range); unit: miles
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 878 | 446
miles | 19.0 [0 to 232] | 18.0 [0 to 240]

18. Secondary Outcome: Intervals in Screening for Diabetic Retinopathy (ISDR) Questionnaire, Time Spent on Visit/Helping on Visit
Description: as for outcome 16
Time Frame: Baseline
Population: ITT. All randomised subjects.
Measure: Median (Full Range); unit: Hours
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
Hours
  Time spent on visit: number analyzed (Participants) | 991 | 496
  Time spent on visit | 2.00 [0.0 to 6.3] | 2.00 [0.0 to 6.0]
  Total time spent helping on visit: number analyzed (Participants) | 393 | 188
  Total time spent helping on visit | 2.00 [0.0 to 6.3] | 2.00 [0.0 to 10.5]

19. Secondary Outcome: Intervals in Screening for Diabetic Retinopathy (ISDR) Questionnaire, Participants/Others Who Took Time Off Work to Attend Visits
Description: as for outcome 16
Time Frame: Baseline
Population: ITT. All randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1027 | 511
Participants
  In employment, YES: number analyzed (Participants) | 1019 | 508
  In employment, YES | 152 | 57
  Took time off work to attend, YES: number analyzed (Participants) | 152 | 57
  Took time off work to attend, YES | 70 | 26
  Assistance by others to attend visit, YES: number analyzed (Participants) | 1013 | 508
  Assistance by others to attend visit, YES | 410 | 197
  Others took time off work to attend, YES: number analyzed (Participants) | 407 | 197
  Others took time off work to attend, YES | 82 | 40

20. Secondary Outcome: Health Care Resource Use Questionnaire
Description: Pharmacoeconomics
  Resources used by the health care staff (per administration), measured by the health care resource use questionnaire.
  The questionnaire assessed the time used by the health care staff during administration of the investigational product and the administration time (including the observational time). The health care participants included in the evaluation were: investigator, pharmacist, physician, study coordinator, study nurse.
  The data for this endpoint show the responses at baseline for both treatment groups.
  The frequency of drug administration between the 2 treatment groups is different (i.e. up to a factor 5 more frequent in the iron sucrose treatment group).
Time Frame: Baseline
Population: ITT. All randomised subjects.
Measure: Median (Full Range); unit: hours
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Health care staff involved in the iron isomaltoside/ferric derisomaltose treatment group.
  Assessment of the time used by the health care staff during administration of the investigational product and the administration time (including the observational time).
- Iron Sucrose: Health care staff involved in the iron sucrose treatment group.
  Assessment of the time used by the health care staff during administration of the investigational product and the administration time (including the observational time).
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 2345 | 1166
hours
  Time spent per site staff | 1.17 [0.0 to 20.8] | 1.00 [0.0 to 20.1]
  Time spent per subject: number analyzed (Participants) | 1020 | 510
  Time spent per subject | 2.58 [0.5 to 20.8] | 2.33 [0.2 to 20.3]

ADVERSE EVENTS:
Time Frame: From the time a subjects had signed the informed consent form (CRF) and until they had completed the study, all adverse events (AEs) or serious adverse events (SAEs) were reported in the CRF. The actual study duration was 8 weeks (or shorted if the trial was discontinued). Overall, eligible subjects participated in the trial for approximately 10 weeks (including a 14-day screening period).
Description: An AE was described as follows: the nature of the event was described in precise, standard medical terminology (i.e. not necessarily the exact words used by the subject). If known, a specific diagnosis was stated. Furthermore, the Investigator described an AE regarding seriousness, severity, relatedness, and outcome.
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
All-Cause Mortality (participants affected / at risk) | 3/1019 | 3/506
Serious Adverse Events (participants affected / at risk) | 83/1019 | 50/506
Other Adverse Events (participants affected / at risk) | 56/1019 | 34/506
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside/Ferric Derisomaltose (N=1019) | Iron Sucrose (N=506)
Cardiac failure congestive (Cardiac disorders) | 7 (7) | 11 (13)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (7) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 5 (5) | 3 (3)
End stage renal disease (Renal and urinary disorders) | 5 (5) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 3 (3)
Death (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside/Ferric Derisomaltose (N=1019) | Iron Sucrose (N=506)
Urinary tract infection (Infections and infestations) | 22 (22) | 14 (14)
Hypertension (Vascular disorders) | 14 (15) | 13 (18)
Hyperkalaemia (Metabolism and nutrition disorders) | 22 (22) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the study results. Before submission for publication or presentation, Institution shall allow Sponsor not less than 90 days to review any manuscript and not less than 30 days to review any poster presentation, abstract, or any other written or oral material which describes or discloses the study results. If sponsor so requests in writing, Institution shall withhold any publication or presentation for an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT02940860/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT02940860/SAP_001.pdf